CLINICAL TRIAL: NCT00688415
Title: A Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacology of VTX-2337 When Administered to Adult Subjects With Advanced Solid Tumors or Lymphoma
Brief Title: Safety and Pharmacologic Study of VTX-2337 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VRXP-A101
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Advanced Solid Tumors; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — VTX-2337

INTERVENTIONS:
Drug: VTX-2337 — Escalating doses of the investigational drug will be administered to cohorts of patients until the highest tolerated dose is identified.

SUMMARY:
This is a multi-center, Phase I study of a new investigational drug, VTX-2337, that may stimulate the immune system to help fight cancer. The purpose of the study is to assess the safety of the investigational drug and to identify the highest dose that is well-tolerated. The pharmacology of VTX-2337 will also be evaluated.

ELIGIBILITY:
Other specific eligibility criteria may apply. Examination by the investigator is necessary to fully determine eligibility.

Inclusion Criteria:

* Ability and willingness to provide written informed consent
* Histologically or cytologically confirmed solid tumors or lymphoma
* Locally advanced or metastatic disease
* Life expectancy of at least 16 weeks
* ECOG performance status of 0 or 1
* Acceptable physical exam and laboratory tests at study entry
* Willingness to use medically acceptable contraception
* A negative serum pregnancy test for women with reproductive potential

Exclusion Criteria:

* Anticancer therapy within 2 weeks
* Treatment with an investigational agent within 4 weeks
* Systemic corticosteroids within 2 weeks or a requirement for systemic immunosuppressive therapy
* Known brain metastases unless stable for at least 28 days
* Active autoimmune disease
* Insulin-dependent diabetes mellitus
* Clinically significant cardiac disease within 6 months
* Significant infection or fever within 1 week
* Pregnant or breast-feeding females
* Other conditions or circumstances that could interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11-07 (Actual); Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and identification of dose-limiting toxicities | Study duration
Pharmacokinetics | First dose of investigational drug

SECONDARY OUTCOMES:
Pharmacodynamics | Study duration
Identification of the MTD | First cycle of investigational drug

CONTACTS AND LOCATIONS:
Overall Officials: Amar Patel, MD, Study Director — Celgene
Locations (2):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona